CLINICAL TRIAL: NCT06914128
Title: A First-in-human Study to Evaluate the Safety, Tolerability and Pharmacokinetics, Pharmacodynamics and Preliminary Clinical Activity of BAY 3713372, a Novel 2nd Generation PRMT5 Inhibitor, in Participants With MTAP-deleted Solid Tumors.
Brief Title: A First-in-human Study to Learn How Safe BAY 3713372 is and How it Works in Participants With MTAP-deleted Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22931; 2025-520623-24-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: MTAP-deleted Solid Tumors
Keywords: Solid Tumors; Non-small cell lung cancer; NSCLC; Pancreatic adenocarcinoma; PDAC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation (Intervention Cohort 1) (Experimental): For the escalation part, different dose levels of BAY 3713372 administered as monotherapy are planned.
  Interventions: Drug: BAY 3713372
- Backfill cohorts in Intervention Cohort 1 (Dose Escalation) (Experimental): Backfill cohorts may be initiated concurrently with dose escalation cohorts to generate additional safety, pharmacokinetic, and pharmacodynamic data to facilitate the selection of the optimal doses for use in further development.
  Interventions: Drug: BAY 3713372
- Dose Expansion (Intervention Cohort 1) (Experimental): Dose expansion with BAY 3713372 monotherapy in selected participants with MTAP-deleted solid tumors.
  Interventions: Drug: BAY 3713372
- Dose Expansion (Intervention Cohort 2) (Experimental): Dose expansion with BAY 3713372 monotherapy in participants with MTAP-deleted non-small cell lung cancer (NSCLC).
  Interventions: Drug: BAY 3713372
- Dose Expansion (Intervention Cohort 3) (Experimental): Dose expansion with BAY 3713372 in combination with other treatments in participants with MTAP-deleted NSCLC.
  Interventions: Drug: BAY 3713372
- Dose Expansion (Intervention Cohort 4) (Experimental): Dose expansion with BAY 3713372 in combination with other treatments in participants with MTAP-deleted NSCLC.
  Interventions: Drug: BAY 3713372
- Dose Expansion (Intervention Cohort 5) (Experimental): Dose expansion with BAY 3713372 monotherapy in participants with MTAP-deleted pancreatic ductal adenocarcinoma (PDAC).
  Interventions: Drug: BAY 3713372
- Dose Expansion (Intervention Cohort 6) (Experimental): Dose expansion with BAY 3713372 in combination with other treatments in participants with MTAP-deleted PDAC.
  Interventions: Drug: BAY 3713372

INTERVENTIONS:
Drug: BAY 3713372 — Daily oral administration

SUMMARY:
The study treatment, BAY 3713372, is under development to treat MTAP (methylthioadenosine phosphorylase)-deleted solid tumors. It is thought to work by blocking the protein arginine N-methyltransferase 5 (PRMT5). This may kill the MTAP-deleted cancer cells while sparing the normal cells.

The main objective of this first-in-human study is to learn how safe BAY 3713372 is, how the body processes it, and how well it works in people with MTAP-deleted solid tumors.

For this, the researchers will study and analyze:

* the number of participants who have adverse events (AEs) after receiving different doses of BAY 3713372 and the AE's severity.
* the number of participants who experience dose-limiting toxicities (DLTs) after receiving different doses of BAY 3713372, the DLT's severity and how often they happened. A DLT is a pre-defined medical problem caused by a specific dose of a drug that is too severe to continue using that dose.
* the total amount of BAY 3713372 in participants' blood (also called AUC) over time after single and multiple doses.
* the highest level of BAY 3713372 in participants' blood (also called Cmax) after single and multiple doses.

Other than the main objective, researchers will also check for the number of participants who show a response to treatment and how long they live without the cancer getting worse.

The study participants will take part in one of the seven distinct groups or "intervention cohorts" of the study. The study will start with a dose escalation phase where distinct groups of participants will receive different doses of BAY 3713372 alone to find the dose that is deemed safe and works best for the participants. When this dose has been found, a larger number of participants will receive BAY 3713372 alone or with other treatments in a dose expansion phase.

Participants may take the study treatment as long as they benefit from the treatment without any severe medical problems.

Participants will visit the study site:

* at least twice before the treatment starts
* multiple times when they start taking the treatment
* once after 30 days of receiving the last dose and every 9 weeks after that until the cancer worsens, or the participant stops for any other reason

During the study, the doctors and their study team will:

* check participants' health by performing tests such as blood and urine tests, and checking heart health using an electrocardiogram
* check if the participants' cancer has grown and/or spread using computed tomography (CT) or magnetic resonance imaging (MRI) and, if needed, bone scan
* take tumor samples

The study doctors and their team will contact the participants every 3 months until 2 years after the last participant's last dose or the end of the study to learn about the participant's health.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years old of age, or the legal age of consent in the jurisdiction of the country in which the study takes place, at the time of signing the informed consent.
* At least one measurable lesion that would qualify as target lesion by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1).
* Homozygous MTAP-deletion identified through molecular testing from a locally certified laboratory.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Previous additional cancer else than the one evaluated in this study within the past 2 years except for basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, superficial bladder tumors, localized prostate cancer or other tumors that in the opinion of the investigator, are considered cured or not immediately life-threatening, and will not interfere with the scientific goals of this study.
* A marked prolongation of QT/QTc interval at screening (e.g., repeated demonstration of a QTc interval >450 ms). Participants with permanent pacemakers (i.e., a paced rhythm) may be eligible based on the investigator's clinical assessment and discretion.
* Cardiac history comprising:

  * History of congestive heart failure Class >II according to the New York Heart Association Functional Classification.
  * Myocardial infarction less than 6 months before the start of study intervention.
  * Serious cardiac arrhythmias requiring treatment or any clinically important abnormalities in rhythm, conduction or morphology on resting ECG with the exception of atrial fibrillation which is well-controlled and requires only digoxin or beta blockers.
* Unstable angina within 4 weeks before start of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2029-06-17 (Estimated); Study Completion 2029-06-17 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation (Master and Intervention Cohort 1): Number of participants with treatment-emergent adverse events (TEAEs) | From the first administration of study intervention up to 30 days after the last dose of study intervention
  TEAEs will be graded according to NCI-CTCAE v.5.0 and will be reported using the latest version of MedDRA coding dictionary
Dose Escalation (Master and Intervention Cohort 1): Number of participants with treatment-emergent serious adverse events (TESAEs) | From the first administration of study intervention up to 30 days after the last dose of study intervention
  TESAEs will be graded according to NCI-CTCAE v.5.0 and will be reported using the latest version of MedDRA coding dictionary
Dose Escalation (Master and Intervention Cohort 1): Severity of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs) | From the first administration of study intervention up to 30 days after the last dose of study intervention
  TEAEs and TESAEs will be graded according to NCI-CTCAE v.5.0 and will be reported using the latest version of MedDRA coding dictionary
Dose Escalation (Master and Intervention Cohort 1): Incidence of dose-limiting toxicities (DLTs) | From the first dose of study intervention to the end of Cycle 1 (each cycle is 21 days)
  DLTs per participants. DLTs will be graded according to NCI-CTCAE v.5.0
Dose Escalation (Master and Intervention Cohort 1): Number of participants with DLTs | From the first dose of study intervention to the end of Cycle 1 (each cycle is 21 days)
  Number of participants with at least one DLT
Dose Escalation (Master and Intervention Cohort 1): Maximum concentration (Cmax) of the respective dosing interval of BAY 3713372 | From the first dose of study intervention up to Cycle 2 Day 1 (each cycle is 21 days)
Dose Escalation (Master and Intervention Cohort 1): Area under the curve (AUC) of the respective dosing interval of BAY 3713372 | From the first dose of study intervention up to Cycle 2 Day 1 (each cycle is 21 days)
Dose Expansion (Master, Intervention Cohorts 1 - 6): Objective response rate (ORR) | Approximately 1.5 years
  Determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Dose Expansion (Intervention Cohorts 3, 4 and 6): Number of participants with DLTs | From the first dose of study intervention to the end of Cycle 1 (each cycle is 21 days, except for Intervention Cohort 6, which has a cycle length of 28 days)
  Number of participants with at least one DLT

SECONDARY OUTCOMES:
Dose Escalation (Master and Intervention Cohort 1): Objective response rate (ORR) | Approximately 1.5 years
  Determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Dose Escalation (Master and Intervention Cohort 1): Duration of response (DOR) | Approximately 3 years
  Determined by the investigator according to RECIST v1.1
Dose Escalation (Master and Intervention Cohort 1): Progression-free survival (PFS) | Approximately 3 years
  Determined by the investigator according to RECIST v1.1
Dose Escalation (Master and Intervention Cohort 1): Time to response (TTR) | Approximately 1.5 years
Dose Expansion (Master, Intervention Cohorts 1 - 6): Number of participants with treatment-emergent adverse events (TEAEs) | From the first administration of study intervention up to 30 days after the last dose of study intervention
  TEAEs will be graded according to NCI-CTCAE v.5.0 and will be reported using the latest version of MedDRA coding dictionary
Dose Expansion (Master, Intervention Cohorts 1 - 6): Number of participants with treatment-emergent serious adverse events (TESAEs) | From the first administration of study intervention up to 30 days after the last dose of study intervention
  TESAEs will be graded according to NCI-CTCAE v.5.0 and will be reported using the latest version of MedDRA coding dictionary
Dose Expansion (Master, Intervention Cohorts 1 - 6): Severity of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs) | From the first administration of study intervention up to 30 days after the last dose of study intervention
  TEAEs and TESAEs will be graded according to NCI-CTCAE v.5.0 and will be reported using the latest version of MedDRA coding dictionary
Dose Expansion (Master, Intervention Cohorts 1, 3, 4, and 6): Incidence of dose-limiting toxicities (DLTs) | From the first dose of study intervention to the end of Cycle 1 (each cycle is 21 days, except for Intervention Cohort 6, which has a cycle length of 28 days)
  DLTs per participants. DLTs will be graded according to NCI-CTCAE v.5.0
Dose Expansion (Master, Intervention Cohorts 1 - 6): Duration of response (DOR) | Approximately 3 years
  Determined by the investigator according to RECIST v1.1
Dose Expansion (Master, Intervention Cohorts 1 - 6): Progression-free survival (PFS) | Approximately 3 years
  Determined by the investigator according to RECIST v1.1
Dose Expansion (Master, Intervention Cohorts 1 - 6): Time to response (TTR) | Approximately 1.5 years
Dose Expansion (Master, Intervention Cohorts 1 - 4, and 6): Maximum concentration (Cmax) of the respective dosing interval of BAY 3713372 | From the first dose of study intervention up to Cycle 2 Day 1 (each cycle is 21 days, except for Intervention Cohort 6, which has a cycle length of 28 days)
Dose Expansion (Master, Intervention Cohorts 1 - 4, and 6): Area under the curve (AUC) of the respective dosing interval of BAY 3713372 | From the first dose of study intervention up to Cycle 2 Day 1 (each cycle is 21 days, except for Intervention Cohort 6, which has a cycle length of 28 days)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (12):
  - UCLA Health Bowyer Oncology Center, Los Angeles, California
  - UCSF Helen Diller Medical Center at Parnassus Heights - Neurology, San Francisco, California
  - Stanford University Medical Center - Neurology, Stanford, California
  - Sarah Cannon Research Institute at HCA HealthONE Presbyterian St. Luke's, Denver, Colorado
  - Sarah Cannon Research Institute at Florida Cancer Specialists- Lake Nona, Orlando, Florida
  - Massachusetts General Hospital - Neurology, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Oncology Department, Boston, Massachusetts
  - START | Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center New York - Main Campus, New York, New York
  - SCRI Oncology Partners, Nashville, Tennessee
  - NEXT Dallas - Oncology Department, Irving, Texas
  - START | San Antonio, San Antonio, Texas
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Concord Repatriation General Hospital (CRGH) (Concord Hospital) - Concord Cancer Centre, Concord, New South Wales
  - Northern Hospital, Epping, New South Wales
  - Calvary Mater Hospital Newcastle - Oncology, Waratah, New South Wales
- Belgium (4):
  - UZ Leuven Gasthuisberg - Pneumology Department, Leuven, Vlaams-Brabant
  - Antwerp University Hospital | Oncology Department, Antwerp
  - Ghent University Hospital | Drug Research Unit Department, Ghent
  - Centre Hospitalier Universitaire (CHU) de Liege - Domaine Universitaire du Sart Tilman - Medical Oncology, Liège
- China (2):
  - Beijing Cancer Hospital - Oncology Department, Beijing, Beijing Municipality
  - Tongji Hosp. of Tongji Med Coll, Huazhong Uni of Sci & Tech., Wuhan, Hubei
- Czechia (2):
  - Masarykova Univerzita - Masarykuv Onkologicky Ustav (MOU) - Klinika Komplexni Onkologicke Pece (KKOP), Brno
  - Fakultní nemocnice Olomouc - Onkologická klinika, Olomouc
- Denmark (2):
  - Rigshospitalet - Kræftbehandling, Copenhagen OE
  - Odense University Hospital - Oncology Department, Odense C
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori - S. C. Oncologia Medica 1, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Fase I, Roma
  - Humanitas Mirasole S.p.A. - Oncologia Medica ed Ematologia, Rozzano
- Japan (4):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shizuoka Cancer Center, Sunto, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- Netherlands (3):
  - Nederlands Kanker Instituut, Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG) - UMC Groningen Comprehensive Cancer Center, Groningen
  - Erasmus Medisch Centrum, Rotterdam
- Singapore (3):
  - National University Hospital Medical Centre, Singapore
  - National Cancer Center Singapore - Oncology Department, Singapore
  - Icon Cancer Centre, Singapore
- Spain (8):
  - Hospital San Pedro | Oncologia, Logroño, La Rioja
  - NEXT - Hospital Universitario Quironsalud Madrid | Oncologia, Pozuelo de Alarcón, Madrid
  - Hospital Hm Nou Delfos | Oncologia, Barcelona
  - Hospital Universitari Vall D Hebron | Oncologia, Barcelona
  - Clinica Universidad De Navarra | Oncologia, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz | Oncologia, Madrid
  - Hospital Universitario Virgen De La Victoria | Oncologia, Málaga
  - Hospital Clinico Universitario De Valencia | Oncologia, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset - Klinisk prövningsenhet Fas I/FIH, Gothenburg
  - Karolinska Universitetssjukhuset - Fas I-enheten Solna CKC, Stockholm
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust | Sutton - Oak Foundation Drug Development Unit, London, Greater London
  - The Christie NHS Foundation Trust | Christie Hospital - Experimental Cancer Medicine Team, Manchester

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.